CLINICAL TRIAL: NCT01530009
Title: The Effect of Amoxicillin Versus Placebo on Gastrointestinal Motility in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Carlo Di Lorenzo, Pediatric Gastroenterologist, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB11-00740
Record Dates: First submitted 2012-02-07; First posted 2012-02-09 (Estimated); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Functional Gastrointestinal Disorders
Keywords: Antroduodenal manometry; Child; Adolescent; Amoxicillin; Gastrointestinal Motility
MeSH Terms: conditions — Gastrointestinal Diseases | interventions — Amoxicillin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amoxicillin (Active Comparator): A liquid preparation of amoxicillin will be administered during the study through a nasoduodenal catheter after random patient assignment.
  Interventions: Drug: Amoxicillin
- Placebo (Placebo Comparator): A liquid placebo will be administered via a nasoduodenal catheter to patients based on random assignment.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Amoxicillin — A liquid preparation of amoxicillin will be administered via a nasoduodenal catheter as a one time dose of 20 mg/kg.
  Other Names: Amoxil; Amoxicot; DisperMox; Moxilin; Trimox; Moxatag
  Arms: Amoxicillin
Other: Placebo — A liquid placebo will be administered via nasoduodenal catheter to patients based on random assignment.
  Arms: Placebo

SUMMARY:
The goal of this study is to determine whether amoxicillin (AMX) alone has an appreciable effect on upper gastrointestinal motility compared to placebo. In particular, induction of phase III of the interdigestive migrating motor complex (MMC) by AMX will be the primary outcome of the study. MMCs are periodic waves of electrical activity resulting in muscular contractions that pass through the walls of the stomach and intestinal tract during the fasting state. It is characterized by an initial period where there is a minimal electrical activity and muscular contraction (phase I), followed by a gradual increase in the frequency of contractions (phase III) that often leads to a characteristic cluster of contractions (phase III). This cycle occurs only in the fasting state in normal individuals and the frequency of phase III is quite varied, dependent on age and the presence of any underlying abnormalities in gastrointestinal motility. Secondary outcomes will include characteristics of the MMC, patient demographics in responders and non-responders, and the safety profile of AMX at the intervention dose.

DETAILED DESCRIPTION:
Motility disorders are common in childhood and can present with a variety of symptoms including recurrent vomiting, abdominal pain and distension. They are often the reason for multiple medical visits and can be associated with significantly impaired quality of life in severe cases. There are a limited number of available medications used to improve motility in the stomach and small bowel, which include dopamine-receptor antagonists, serotonergic agents and antibiotics such as erythromycin. Among the latter group, amoxicillin-clavulanate (AMC) has been shown to enhance fasting small intestinal motility in adults and children. The mechanism of action is not currently known though theories include indirect release of an intraluminal mediator such as motilin, or direct interaction of the β-lactam moiety with γ-aminobutyric acid receptors in the myenteric plexus.

AMC is a combination of amoxicillin (AMX) with clavulanic acid (CA), a β-lactamase inhibitor. This modification of the drug results in a broader spectrum of antibacterial activity to include AMX sensitive and β-lactamase-producing strains. Although both AMX and AMC are generally well tolerated, AMX can be associated with fewer adverse effects due to the presence of the CA moiety in AMC. AMC is associated with a higher frequency of nausea, vomiting and transient diarrhea compared to AMX. In a study of outpatient children, patients on AMC have been shown to have an increased risk of antibiotic-associated diarrhea. Drug-related liver injury is also more common in patients taking AMC. Furthermore, it is advisable to use the most narrow spectrum antibiotic that demonstrates clinical efficacy in light of the emergence of β-lactam-β-lactamase inhibitor-resistant bacterial strains accelerated by excess antibiotic use.

AMX has a good safety profile and is frequently prescribed for children by community physicians based on history and physical examination alone. It is the recommended first line treatment in common childhood illnesses such as upper respiratory infections, including ear and sinus infections, and community-acquired pneumonia.

The goal of this study is to determine whether a single dose of AMX has an appreciable effect on upper gastrointestinal motility compared to placebo. In particular, induction of phase III of the interdigestive migrating motor complex (MMC) by AMX will be the primary outcome of the study. MMCs are periodic waves of electrical activity resulting in muscular contractions that pass through the walls of the stomach and intestinal tract during the fasting state. It is characterized by an initial period where there is a minimal electrical activity and muscular contraction (phase I), followed by a gradual increase in the frequency of contractions (phase III) that often leads to a characteristic cluster of contractions (phase III). This cycle occurs only in the fasting state in normal individuals and the frequency of phase III is quite varied, dependent on age and the presence of any underlying abnormalities in gastrointestinal motility. Secondary outcomes will include characteristics of the MMC, patient demographics in responders and non-responders, and the safety profile of AMX at the intervention dose.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3-21 years referred to the Motility Department at Nationwide Children's Hospital for antroduodenal manometry testing

Exclusion Criteria:

* History of allergic reaction to amoxicillin, amoxicillin-clavulanate, or cephalosporins with a common-side chain (e.g. cefadroxil, cefprozil, cefatrizine)
* Therapy with a prokinetic within 3 days of the scheduled antroduodenal manometry
* Families who do not agree to participate

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2022-01 (Actual); Study Completion 2022-01 (Actual)

PRIMARY OUTCOMES:
Induction of phase III of the migrating motor complex | 30 minutes after study drug administration
  The migrating motor complex passes through the GI tract during fasting. It is initially characterized by minimal electrical activity and muscular contraction (phase I), followed by an increase in the frequency of contractions (phase III) and finally a characteristic cluster of contractions (phase III). This cycle occurs only in the fasting state in normal individuals and the frequency of phase III depends on age and the presence of any underlying gastrointestinal dysmotility. The primary outcome is to determine whether amoxicillin can induce phase III of the MMC.

SECONDARY OUTCOMES:
Characteristics of the induced phase III of the migrating motor complex | Within 6 months after study drug administration during data analysis phase of study
  Characteristics of the induced phase III of the migrating motor complex will be analyzed.
Patient demographics | Within 6 months after study drug administration during data analysis phase of study
  Patient demographics including age, gender, symptoms and underlying diagnosis will be analyzed in both study groups and compared.
Adverse events after study drug administration | Within 4 hours of study drug administration
  Any adverse events within 4 hours of study drug administration will be recorded and analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Di Lorenzo, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No